CLINICAL TRIAL: NCT06522269
Title: Emergency Stroke Unit for Acute Cerebrovascular Events--A Prospective, Multicenter, Week-wise Randomized, Controlled Trial ( ESU-ACE-C )
Brief Title: Emergency Stroke Unit for Acute Cerebrovascular Events ( ESU-ACE-C )
Status: Completed | Phase: Phase 3 | Type: Interventional
Sponsor: Beijing Tiantan Hospital (Other)
Responsible Party: Principal Investigator, Yongjun Wang, professor, Beijing Tiantan Hospital
Allocation: Randomized | Model: Parallel | Masking: Single | Purpose: Treatment
Other Study IDs: KY2024-131-02-C
Record Dates: First submitted 2024-06-26; First posted 2024-07-26 (Actual); Last update posted 2025-08-22 (Actual); Status verified 2024-08

CONDITIONS: Ischemic Stroke, Acute
Keywords: Emergency stroke unit; Low-field magnetic resonance imaging; Reperfusion therapy
MeSH Terms: conditions — Ischemic Stroke

STUDY DESIGN:
Who Masked: Outcomes Assessor
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No | US Export: No

ARMS (2):
- Emergency Stroke Unit based on 0.23-T MRI (Experimental): The participants with hyperacute ischemic stroke (arriving at the emergency department within 4.5 hours of symptom onset) who are eligible to receive reperfusion therapy will be managed by Emergency Stroke Unit process based on low-field magnetic resonance imaging.
  Interventions: Combination Product: Emergency Stroke Unit based on 0.23-T MRI
- Standard stroke unit adherent to guidelines (Placebo Comparator): The participants with hyperacute ischemic stroke (arriving at the emergency department within 4.5 hours of symptom onset) who are eligible to receive reperfusion therapy will be managed by standard stroke unit process adherent to guidelines.
  Interventions: Combination Product: Standard stroke unit adherent to guidelines

INTERVENTIONS:
Combination Product: Emergency Stroke Unit based on 0.23-T MRI — The participants with hyperacute ischemic stroke (arriving at the emergency department within 4.5 hours of symptom onset) who are eligible to receive reperfusion therapy will be managed by Emergency Stroke Unit process based on low-field magnetic resonance imaging.
  Arms: Emergency Stroke Unit based on 0.23-T MRI
Combination Product: Standard stroke unit adherent to guidelines — The participants with hyperacute ischemic stroke (arriving at the emergency department within 4.5 hours of symptom onset) who are eligible to receive reperfusion therapy will be managed by standard stroke unit process adherent to guidelines.
  Arms: Standard stroke unit adherent to guidelines

SUMMARY:
To compare the prognosis of patients with hyperacute ischemic stroke (who arrive at the emergency department within 4.5 hours of symptom onset) managed in a standard stroke unit adherent to guidelines versus managed in Emergency Stroke Unit (a new stroke unit based on low-field magnetic resonance imaging).

DETAILED DESCRIPTION:
The first MRI machines in the 1970s and 1980s were low-field due to technological limitations. As technology advanced, the focus shifted to higher field strengths to achieve better image resolution and faster scan times. Recently, there has been renewed interest in low-field MRI due to advancements in hardware and software, making them more viable for specific clinical applications, including acute stroke. Prompt and accurate imaging is crucial for diagnosing ischemic stroke and determining the appropriate treatment (e.g., thrombolysis or thrombectomy). Research has demonstrated that low-field MRI can effectively detect acute ischemic changes and distinguish between ischemic and hemorrhagic stroke. By providing accessible, cost-effective, and safe imaging, it can facilitate timely and accurate treatment, particularly in settings where high-field MRI is not readily available. This prospective, multicenter, week-wise randomized controlled trial will compare the prognosis of patients with hyperacute ischemic stroke (who arrive at the emergency department within 4.5 hours of symptom onset) managed in a standard stroke unit adherent to guidelines versus managed in Emergency Stroke Unit (a new stroke unit based on low-field magnetic resonance imaging).

ELIGIBILITY:
Inclusion Criteria:

1. Age ≥ 18 years;
2. Patients who arrive at the emergency department within 4.5 hours of symptom onset* (*Symptom onset is defined by the "last seen normal" principle);
3. Presenting with ischemic stroke symptoms;
4. Pre-stroke mRS score 0-1;
5. Baseline NIHSS score ≥ 5;
6. Eligible for rt-PA/TNK thrombolysis;
7. Informed consent signed.

Exclusion Criteria:

1. Baseline NIHSS score < 5;
2. Unable to undergo MRI because of claustrophobia;
3. Patients with cardiac pacemaker/brain pacemaker/insulin pump implantation;
4. Definite contraindication for rt-PA/TNK thrombolysis;
5. Patients with postictal hemiparesis (Todd's paralysis) or those with concomitant neurological/psychiatric conditions who are unable or unwilling to cooperate;
6. Pregnant women, nursing mothers, or reluctance to use effective contraceptive measures during the period of trial;
7. Participation in other interventional randomized clinical trials within 3 months before enrollment;
8. Patients deemed unsuitable for participation in this trial by the investigator or those for whom participation in this trial may result in greater risks.

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 1622 (Actual)
Dates: Start 2024-08-08 (Actual); Primary Completion 2025-08-15 (Actual); Study Completion 2025-08-15 (Actual)

PRIMARY OUTCOMES:
The utility-weighted modified Rankin Scale (uw-mRS) at 90 days (± 7 days). | at 90 days (± 7 days)
  The utility-weighted modified Rankin Scale (uw-mRS) at 90 days (± 7 days). Scores on the modified Rankin scale range from 0 (no neurologic deficit) to 6 (death).

SECONDARY OUTCOMES:
Ordinal (shift) analysis of modified Rankin Scale (mRS) at 90 days (± 7 days). | at 90 days (± 7 days)
  Ordinal (shift) analysis of modified Rankin Scale (mRS) at 90 days (± 7 days). Scores on the modified Rankin scale range from 0 (no neurologic deficit) to 6 (death).
Excellent functional outcome (Modified Rankin Scale score, mRS 0-1) at 90 days (± 7 days). | at 90 days (± 7 days)
  Excellent functional outcome (Modified Rankin Scale score, mRS 0-1) at 90 days (± 7 days). Scores on the modified Rankin scale range from 0 (no neurologic deficit) to 6 (death).
Good functional outcome (Modified Rankin Scale score, mRS 0-2) at 90 days (± 7 days). | at 90 days (± 7 days)
  Good functional outcome (Modified Rankin Scale score, mRS 0-2) at 90 days (± 7 days). Scores on the modified Rankin scale range from 0 (no neurologic deficit) to 6 (death).
A 30% reduction (improvement) from baseline to 24 hours in the NIHSS score. | from baseline to 24 hours in the NIHSS score.
  A 30% reduction (improvement) from baseline to 24 hours in the NIHSS score. Scores on the National Institutes of Health Stroke Scale (NIHSS) range from 0 to 42, with higher scores indicating greater neurological deficits.
The time from symptoms onset to intravenous thrombolysis decision. | up to 4.5 hours from symptom onset
  The time from symptoms onset to intravenous thrombolysis decision.
The time from emergency department arrival to intravenous thrombolysis decision. | up to 4.5 hours from symptom onset.
  The time from emergency department arrival to intravenous thrombolysis decision.
Proportion of participants ultimately treated with reperfusion therapy (separated rate of intravenous thrombolysis / endovascular thrombectomy / bridging therapy). | up to 6 hours from symptom onset.
  Proportion of participants ultimately treated with reperfusion therapy (separated rate of intravenous thrombolysis / endovascular thrombectomy [within 6 hours from symptom onset / all patients] / bridging therapy).
The time from emergency department arrival to the start of intravenous thrombolysis. | up to 4.5 hours from symptom onset
  The time from emergency department arrival to the start of intravenous thrombolysis.
The cost-effectiveness analysis. | up to 3 months from enrollment.
  Cost Effectiveness as measured by average patient QALYs, post-stroke healthcare utilization, incremental fixed costs associated with the ESU.
Symptomatic intracranial hemorrhages (according to the ECASS III criteria) within 36 hours. | within 36 hours.
  Symptomatic intracranial hemorrhages within 36 hours (sICH definition: according to the ECASS III criteria: any apparently extravascular blood in the brain or within the cranium that was associated with clinical deterioration, as defined by an increase of 4 points or more in the score on the NIHSS, or that led to death and that was identified as the predominant cause of the neurological deterioration).
Symptomatic intracranial hemorrhages (according to the ECASS III criteria) at 90 days (± 7 days). | at 90 days (± 7 days).
  Symptomatic intracranial hemorrhages at 90 days (± 7 days) (sICH definition: according to the ECASS III criteria: any apparently extravascular blood in the brain or within the cranium that was associated with clinical deterioration, as defined by an increase of 4 points or more in the score on the NIHSS, or that led to death and that was identified as the predominant cause of the neurological deterioration).
Mortality at 90 days (± 7 days). | at 90 days (± 7 days).
Adverse events at 90 days (± 7 days). | at 90 days (± 7 days).
Serious adverse events at 90 days (± 7 days). | at 90 days (± 7 days).

CONTACTS AND LOCATIONS:
Overall Officials: Yongjun Wang, Study Director — Beijing Tiantan Hospital
Locations (1):
- Beijing Tiantan Hospital, Capital Medical University, Beijing, China

IPD SHARING:
Plan to Share IPD: No